CLINICAL TRIAL: NCT01331213
Title: Effect of Pregabalin on Colonic Motor and Sensory Function in Adults With Irritable Bowel Syndrome With Predominant Constipation
Brief Title: Pregabalin on Colonic Motor and Sensory Function in Constipation Predominant Irritable Bowel Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Michael Camilleri, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 11-000485; UL1RR024150 (NIH)
Record Dates: First submitted 2011-04-06; First posted 2011-04-07 (Estimated); Results first posted 2014-03-03 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-01

CONDITIONS: Irritable Bowel Syndrome
Keywords: Pregabalin; Irritable Bowel Syndrome; motor; sensation; colon; human
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pregabalin (Active Comparator): Subjects randomized to this arm received a single dose of pregabalin 200mg orally.
  Interventions: Drug: Pregabalin
- Placebo (Placebo Comparator): Subjects randomized to this arm received a single dose of placebo orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — FDA approved medication (capsules) at 200mg dose.
  Other Names: Lyrica
  Arms: Pregabalin
Drug: Placebo — Placebo capsules
  Arms: Placebo

SUMMARY:
The general aim of the current study is to describe the effect of pregabalin on colonic and sensory functions in adults with constipation predominant irritable bowel syndrome (IBS-C).

Study hypotheses:

1. Single-dose pregabalin 200mg increases sensation thresholds and decreases sensation ratings in response to balloon distension in the colon relative to pre-pregabalin treatment.
2. Single-dose pregabalin 200 mg will increase colonic compliance and decrease colonic pain and gas thresholds in patients with irritable bowel syndrome constipation predominant.
3. Single-dose pregabalin 200mg increases the colonic phasic and tonic response to a standardized meal.

DETAILED DESCRIPTION:
The treatment of patients with irritable bowel syndrome and chronic abdominal pain is advancing with several effective options for symptoms related to bowel dysfunction and bloating/distension. However, there are no approved or effective centrally or peripherally acting visceral analgesics. Pregabalin has been proposed as a treatment for visceral pain, based on the pharmacological actions, and efficacy in neuropathic pain.

This was a trial in adults with IBS-C to compare the effects of oral pregabalin 200 mg versus placebo on colon motility, sensation, and tone.

All participants presented on the study day after an overnight bowel preparation with an oral colonic lavage solution and a 12-hour fast. Flexible colonoscopy to the splenic flexure was performed without sedation by one investigator. The barostat catheter (constructed at Mayo Clinic, Rochester, MN) incorporating six manometric point sensors 5 cm apart was introduced into the colon over a guidewire, and the polyethylene balloon (10 cm long, cylindrical shape with a maximum volume of 600 ml) was placed in the mid-descending or junction of the sigmoid and descending colon. A rigid-piston barostat was used to measure intraballoon pressure and volume throughout the study. After an initial inflation to a volume of 75 ml to ensure unfolding of the balloon, the operating pressure was identified as the distension pressure at which respiratory excursions were recorded clearly from the barostat tracing, and the intraballoon pressure was set 2 mm Hg above the minimal distension pressure. A conditioning distention from 0 to 20 mmHg in increments of 2 mmHg every 15 seconds was performed over a period of 75 seconds.

After an equilibration period of 10 minutes, a 100-mm visual analog scale (VAS) was used to assess the level of anxiety or stress experienced by each subject because they are potentially significant covariates in the assessment of visceral sensation scores.

Colonic compliance was assessed by the ascending methods of limit (ramp-like increases of 4 mm Hg at 60-second intervals). During the assessment of colonic compliance, participants reported their thresholds for first perception, gas and pain. After another 10 minute equilibration period, fasting colonic tone was measured at operating pressure for a period of 10 minutes.

Randomized-order phasic distentions were then applied at 16, 24, 30, and 36 mmHg above the operating pressure to measure the sensations of gas and pain. Each distention lasted 1 minute and was followed by an equilibration period at the operating pressure for 2 minutes. A 100-mm visual analog scale (VAS) was used to assess the rating of arousal and stress experienced by each participant before performing the phasic distentions. During the distentions, participants also used the 100-mm VAS to rate the intensity of gas and pain perception at 30 seconds from the start of the distention.

Colonic compliance, fasting tone, pressure thresholds for first perception, gas, and pain, and VAS scores of gas and pain during the phasic distentions were measured before administering the study medication and 1 hour after drug administration. After the postdrug assessment of sensation with phasic distentions, a 30-min assessment of fasting colonic tone was measured in each participant; this provided a baseline to compare the effect of a standard 750-ml chocolate milkshake meal across treatment groups. Postprandial tone was measured over 60 minutes, with the main focus on the first 30 minutes. When the recording was completed, the balloon was deflated and the tube removed by gentle traction.

ELIGIBILITY:
Inclusion criteria:

- Male or females with Constipation Predominant IBS, age 18-65

Exclusion criteria:

* Abdominal surgery other than appendectomy, laparoscopic cholecystectomy, cesarean section, vaginal or laparoscopic hysterectomy or tubal ligation
* Uncontrolled hypertension
* Use of medications that may interact with the study medication
* Use of any of the study medications within the past 30 days
* Pregnancy
* History of chronic renal insufficiency (serum creatinine >1.5mg/dL)
* Psychiatric or psychologic dysfunction
* Current pelvic floor dysfunction
* diagnosis of lactose intolerance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-04; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study between 4/2011 and 3/2012 at the Mayo Clinic in Rochester, Minnesota.
Period: Overall Study
Arm/Group | Pregabalin | Placebo
Started | 8 | 10
Completed | 8 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Placebo | Total
Number analyzed (Participants) | 8 | 10 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (5.88) | 44.1 (11.51) | 44.06 (9.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: Colonic Compliance
Description: Colonic compliance is a measure of the "stiffness" of the colon, that is, what pressure was needed to reach half the maximum volume of the colon. After the barostat balloon catheter was inserted in the mid-descending or junction of the sigmoid and descending colon, the balloon was inflated. After an initial conditioning distension to 20 mm Hg, colonic compliance was measured by step-wise inflation with increments of 4 mm Hg. Colonic compliance was analyzed by a validated linear interpolation method. The pressure at half maximum volume serves as a summary of colonic compliance.
Time Frame: baseline (1 hour before drug administration), post-treatment (1 hour after drug administration)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 8 | 10
mm Hg
  Baseline | 18.96 (4.84) | 16.86 (8.97)
  Post-Treatment | 15.99 (6.4) | 15.75 (7.89)

2. Primary Outcome: Postprandial Colonic Tone [Reported as the Symmetric Percent [Change} in Baseline Colonic Barostat Balloon Volume
Description: The symmetric percent reduction in baseline colonic barostat balloon volume during the first 30 minutes postprandially (PP) corrected for the preprandial (30 min) tone, (symmetric percent change= 100*log_e[fasting/PP]). A positive symmetric percent change reflects a decrease in barostat balloon volume indicating a reduction in colonic tone. (The balloon was placed in the mid-descending or junction of the sigmoid and descending colon.)
Time Frame: The first 30 minutes postprandially, and preprandial (30 minutes)
Measure: Mean (Standard Deviation); unit: Symmetric percentage change
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 8 | 10
Symmetric percentage change | -22.34 (12.98) | -24.45 (12.3)

3. Primary Outcome: Sensory Threshold for Pain
Description: The sensory threshold for first perception of pain was measured by stepwise inflation of the balloon in increments of 4 mm Hg at 60 second intervals. The balloon was placed in the mid-descending or junction of the sigmoid and descending colon. During this assessment participants were asked to report when they had the first perception of pain. The investigator recorded the threshold pressure at which the participants reported this sensation.
Time Frame: approximately 60 minutes after drug administration
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 8 | 10
mm Hg | 36.0 (17.59) | 38.0 (21.02)

4. Primary Outcome: Overall Sensory Ratings in Response to 16, 24, 30 and 36 mm Hg Distensions.
Description: The mm Hg distensions refer to the barostat balloon, which was placed in the mid-descending or junction of the sigmoid and descending colon. Pain sensation was measured by a 100 mm long Visual Analog Scale (VAS). The VAS does not have any pre-set marks between the extremes. For the pain VAS, 0 means no pain and 100 mm means extreme pain. The investigator measures the mark made by the participant in mm and records this for the value of pain.
Time Frame: Approximately 60 minutes after drug administration
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 8 | 10
mm
  Sensation ratings of pain at 16 mm Hg distension | 53.0 (11.83) | 52.3 (20.44)
  Sensation ratings of pain at 24 mm Hg distension | 57.43 (30.49) | 59.60 (26.71)
  Sensation ratings of pain at 30 mm Hg distension | 64.0 (26.12) | 60.3 (24.99)
  Sensation ratings of pain at 36 mm Hg distension | 59.0 (21.93) | 53.7 (33.4)

5. Secondary Outcome: Fasting Colonic Tone
Description: Colonic tone is a measurement of the volume of the colon. Colonic tone was assessed by noting the changes in the balloon volume in the presence of a constant operating pressure in the balloon (in the barostat-manometric assembly placed in the colon.)
Time Frame: Approximately 60 minutes after drug administration
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 8 | 10
mL | 120.4 (12.76) | 116.8 (24.75)

6. Secondary Outcome: Colonic Motility Index
Description: The postprandial motility index (MI)=log_e[number of contractions * sum of amplitudes) + 1] A normal fasting average motility index (MI) would be about 12. An increase in MI means an increase in the phasic contractions (in contrast to tone) which is measured as a change in volume of the barostatically-controlled balloon. (Therefore, an increase in MI means that the meal is moving more quickly through the colon.)
Time Frame: Approximately 1 hour after meal
Measure: Mean (Standard Deviation); unit: log mm Hg
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 8 | 10
log mm Hg
  Post-treatment, descending colon | 13.69 (0.82) | 12.27 (2.09)
  Post-treatment, sigmoid colon | 11.72 (1.58) | 10.21 (3.20)

7. Secondary Outcome: Post-treatment Sensory Threshold for Gas
Description: The sensory threshold for first perception of gas was measured by stepwise inflation of the balloon in increments of 4 mm Hg at 60 second intervals. The balloon was placed in the mid-descending or junction of the sigmoid and descending colon. During this assessment participants were asked to report when they had the first perception of gas. The investigator recorded the threshold pressure at which the participants reported this sensation.
Time Frame: Approximately 60 minutes after drug administration
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 8 | 10
mm Hg | 24.0 (12.65) | 19.2 (13.31)

ADVERSE EVENTS:
Arm/Group | Pregabalin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/10
Other Adverse Events (participants affected / at risk) | 0/8 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No